CLINICAL TRIAL: NCT05305677
Title: Effect of NMN (Nicotinamide Mononucleotide) Intervention on Patients With Polycystic Ovary Syndrome
Brief Title: Effect of NMN (Nicotinamide Mononucleotide) on Polycystic Ovary Syndrome
Acronym: NMN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: M2021577
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; reproductive endocrine; metabolism; gut microbiota; NMN
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMN intervention (Experimental): 8 weeks of NMN
  Interventions: Dietary Supplement: NMN intervention
- Placebo (Placebo Comparator): 8 weeks of NMN-free placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: NMN intervention — NMN capsules (total of 600mg/day) for 8 weeks
  Arms: NMN intervention
Other: Placebo — NMN-free placebo capsules for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to understand the effect of Nicotinamide mononucleotide (NMN) on patients with polycystic ovary syndrome.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of NMN on reproductive endocrine and metabolism, chronic inflammation, and reproductive outcomes in women with polycystic ovary syndrome (PCOS), and to explore its underlying mechanisms to provide the intervention strategies for PCOS.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are 20 to 40 years old;
2. BMI < 25 kg/m2;
3. Individuals with PCOS should meet all the Rotterdam diagnostic criteria: 1) Oligo- and/or anovulation; 2) Clinical and/or biochemical signs of hyperandrogenism; 3) Polycystic ovaries, and exclusion of other aetiologies (congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome).
4. Individuals who can insist on continuous monitoring in the outpatient clinic.
5. Individuals who are not participating in other research projects currently or 3 months before the intervention.

Exclusion Criteria:

1. Individuals who suffering from other diseases that may cause hyperandrogenism and ovulation abnormalities.
2. Individuals who are during pregnant, lactation or menopause.
3. Individuals who currently receiving weight-loss drugs or surgery or within the past 2 months.
4. Individuals who take niacin, nicotinamide, or other vitamin B-related supplementation currently or within the past 2 months.
5. Individuals who need regular medication to treat chronic diseases such as diabetes, hypertension, gout, hyperuricemia, etc.
6. Use of medications that affect hormone levels, appetite, carbohydrate absorption, and metabolism within the past 2 months.
7. Individuals with severe liver diseases or kidney disease that are ineligible to participate in the study.
8. A medical history of severe cardiovascular and cerebrovascular diseases.
9. Individuals who currently suffer from severe gastrointestinal diseases or undergo gastrointestinal resection that may affect nutrient absorption.
10. Individuals who drink more than 15g of alcohol per day or have a smoking habit.
11. Individuals who need drug treatment for any mental illness such as epilepsy and depression.
12. Cancer patients.
13. Individuals who suffer from infectious diseases such as hepatitis B, active tuberculosis, AIDS, etc.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Testosterone level | From enrollment to the end of treatment at 8 weeks
  Changes of testosterone level in serum after intervention.
Antral follicle counts | From enrollment to the end of treatment at 8 weeks
  The number of antral follicle counts in each ovary will be determined using transvaginal ultrasonography for each participant.
Menstrual cycle | before and after 8 weeks of intervention
  The changes of menstrual cycle frequency after intervention.

SECONDARY OUTCOMES:
Luteinizing hormone (LH) level | From enrollment to the end of treatment at 8 weeks
  Changes of LH level in serum after intervention.
Follicle-stimulating hormone (FSH) level | From enrollment to the end of treatment at 8 weeks
  Changes of FSH level in serum after intervention.
Homeostasis Model Assessment for Insulin Resistance (HOMA-IR) index | From enrollment to the end of treatment at 8 weeks
  Changes in HOMA-IR index (fasting insulin * fasting glucose/22.5) after intervention.
Changes in other endocrine hormones | From enrollment to the end of treatment at 8 weeks
Changes in blood NAD+ level and related metabolites | From enrollment to the end of treatment at 8 weeks
Multi-omics | From enrollment to the end of treatment at 8 weeks
  Collect samples before and after 2, 4, 8 weeks of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Patients' information is requested to be confidential.